CLINICAL TRIAL: NCT00185224
Title: A Single-center, Open-label, Controlled, Randomized Study to Investigate the Impact of a Sequential Oral Contraceptive (SH T00658ID) as Compared to a Sequential Oral Contraceptive Containing Ethinylestradiol and Levonorgestrel (SH D00264A) on Plasma Lipids, Hemostatic Variables, and Carbohydrate Metabolism in Healthy Female Volunteers Aged 18-50 Years Over 7 Treatment Cycles, Including the Pharmacokinetics
Brief Title: Metabolism Study to Investigate the Impact of a Sequential Oral Contraceptive
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Healthcare AG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 90927; EudraCT: 2004-001614-13; 301886
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2011-07

CONDITIONS: Contraception
MeSH Terms: interventions — Ethinyl Estradiol-Norgestrel Combination

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: EV/DNG (Qlaira, BAY86-5027, SH T00658K)
- Arm 2 (Active Comparator)
  Interventions: Drug: SH D00264A (Triquilar)

INTERVENTIONS:
Drug: EV/DNG (Qlaira, BAY86-5027, SH T00658K) — 7 treatment cycles of 28 days each (no tablet-free intervals); Days 1-2: 3.0 mg EV; Days 3-7: 2.0 mg EV + 2.0 mg DNG; Days 8-24: 2.0 mg EV + 3.0 mg DNG; Days 25-26: 1.0 mg EV; Days 27 - 28: Placebo
  Arms: Arm 1
Drug: SH D00264A (Triquilar) — 7 treatment cycles of 28 days each (no tablet-free intervals);Days 1-6: 0.03 mg EE + 0.05 mg LNG; Days 7-11: 0.04 mg EE + 0.075 mg LNG; Days 12-21: 0.03 mg EE + 0.125 mg LNG;Days 22-28: Placebo
  Arms: Arm 2

SUMMARY:
The purpose of this study is to confirm the safety of SH T00658ID with regard to plasma lipids, hemostatic variables, and carbohydrate metabolism. In addition, the pharmacokinetic parameter following the long term administration of SH T00658ID will be assessed.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers between 18 and 50 years requiring contraception

Exclusion Criteria:

* Pregnancy or lactation
* Any conditions that might interfere with the outcome as well as all contraindications for OC use

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2005-03; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Impact on metabolic parameters (e.g. hemostatic parameters) after 6 month treatment | Baseline, Cycle 7

SECONDARY OUTCOMES:
Measurement of PK parameters | Cycle 4, Cycle 7

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Bayer Schering Pharma AG - Clin. Pharm. Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Junge W, Mellinger U, Parke S, Serrani M. Metabolic and haemostatic effects of estradiol valerate/dienogest, a novel oral contraceptive: a randomized, open-label, single-centre study. Clin Drug Investig. 2011;31(8):573-584. doi: 10.2165/11590220-000000000-00000. PMID 21721593